CLINICAL TRIAL: NCT01390194
Title: Rapid 10-Minute Liver MRI Protocol in Patients With Suspected Hepatocellular Carcinoma: A Pilot Study to Assess the Image Quality (Multitransmit Body MRI Program)
Brief Title: Rapid 10-Minute Liver MRI Protocol in Patients With Suspected Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: Philips Medical Systems (Industry); Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 0246-10-FB
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Underlying Liver Disease; Hepatitis; Fibrosis of Liver; Cirrhosis With Suspicion of Liver Cancer; Lesion on a Prior Ultrasound, CT or Outside MRI
Keywords: liver disease; hepatocellular carcinoma
MeSH Terms: conditions — Hepatitis; Liver Cirrhosis; Liver Diseases; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- subjects with an underlying liver disease: (1)underlying liver disease; (2) have a lesion on a prior imaging study; (3) must be prior standard MR

SUMMARY:
The purpose of this study to assess the image quality of the rapid magnetic resonance imaging (MRI) compared to the standard MRI.

DETAILED DESCRIPTION:
This is a pilot study to compare a rapid 10-minute liver magnetic resonance imaging (MRI) protocol to standard MRI in participants with suspected hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. underlying liver disease
2. have a lesion on a prior imaging study
3. must have prior standard MR

Exclusion Criteria:

1. Contra-indication for MR imaging including pacemaker, claustrophobia, pregnancy, electronic or vascular devices that are contraindicated;
2. patients with severe kidney dysfunction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with an underlying liver disease
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
image quality outcome | 2 years
  Two MRI exams will be evaluated by two radiologists based on a number of items.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Hussain, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States